CLINICAL TRIAL: NCT01228331
Title: A Randomized Multi-Center Treatment Study (COALL 08-09) to Improve the Survival of Children with Acute Lymphoblastic Leukemia on Behalf of the German Society of Pediatric Hematology and Oncology
Brief Title: Clofarabine or High-Dose Cytarabine and Pegaspargase in Children with ALL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000686545; 2009-012758-18 (EudraCT Number)
Record Dates: First submitted 2010-10-23; First posted 2010-10-26 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-01

CONDITIONS: Leukemia
Keywords: childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Amsacrine; Clofarabine; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; etoposide phosphate; Mercaptopurine; Methotrexate; Methylprednisolone; pegaspargase; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I intensification (cytarabine) (Active Comparator): LR-S patients receive HD cytarabine IV 4 x 3 g over 12 hours daily on days 29-31 and pegaspargase IV over 2 hours on days 31, 52, and 80.
  LR-I and precursor B-cell ALL HR-S and HR-I patients receive HD cytarabine IV 2.500 over 3 hours twice daily on days 29-31 and 106-108 and pegaspargase IV over 2 hours on days 31, 53, 67, and 108.
  Followed by standard consolidation therapy regarding to stratification containing:
  methotrexate, cyclophosphamide, thioguanin, mercaptopurine, etoposide phosphate, amsacrine, cytarabine, methylprednisolone, dexamethasone, vincristine sulfate; whole-brain radiation therapy only if indicated in patients with cns involvement or T-cell ALL
  Interventions: Drug: Amsacrine; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Etoposide phosphate; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine sulfate; Radiation: Whole-brain radiation therapy
- Arm II intensification (clofarabine) (Active Comparator): LR-S patients receive clofarabine* IV 5 x 40 mg over 2 hours every day on days 29-33 and pegaspargase IV over 2 hours on days 33, 52, and 80.
  LR-I and precursor B-cell ALL HR-S and HR-I patients receive clofarabine* IV over 2 hours on days 29-33 and pegaspargase IV over 2 hours on days 33, 53, 67, and 108.
  Followed by standard consolidation therapy regarding to stratification containing:
  methotrexate, cyclophosphamide, thioguanin, mercaptopurine, etoposide phosphate, amsacrine, cytarabine, methylprednisolone, dexamethasone, vincristine sulfate; whole-brain radiation therapy only if indicated in patients with cns involvement or T-cell ALL
  Interventions: Drug: Amsacrine; Drug: Clofarabine; Drug: Cyclophosphamide; Drug: Daunorubicin hydrochloride; Drug: Dexamethasone; Drug: Etoposide phosphate; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine sulfate; Radiation: Whole-brain radiation therapy
- Arm III reinduct.(doxorubicin hydrochl.) (Active Comparator): LR-S patients receive doxorubicin hydrochloride IV 30 mg/m2 over 24 hours on days 1 and 8.
  LR-I, HR-S and HR-I Patients receive doxorubicin hydrochloride IV 30 mg/m2 over 24 hours on days 1, 8, 22, and 29.
  Followed by standard reinduction and maintenance therapy containing:
  cyclophophamide, cytarabine, thioguanine, mercaptopurine, methotrexate and pegaspargase, dexamethasone, vincristine sulfate
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin hydrochloride; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Vincristine sulfate
- Arm IV reinduct.(daunorubicin hydrochl.) (Active Comparator): LR-S patients receive daunorubicin hydrochloride IV 36 mg/m2 over 24 hours on days 1 and 8.
  LR-I, HR-S and HR-I Patients receive daunorubicin hydrochloride IV 36 mg/m2 over 24 hours on days 1, 8, 22, and 29.
  Followed by standard reinduction and maintenance therapy containing:
  cyclophophamide, cytarabine, thioguanine, mercaptopurine, methotrexate and pegaspargase, dexamethasone, vincristine sulfate
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin hydrochloride; Drug: Dexamethasone; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Vincristine sulfate

INTERVENTIONS:
Drug: Amsacrine — one block amsacrine together with etoposide and methylprednisolone for very high risk patients
  Arms: Arm I intensification (cytarabine); Arm II intensification (clofarabine)
Drug: Clofarabine — one block clofarabine with Asparaginase for MRD positive patients after induction
  Arms: Arm II intensification (clofarabine)
Drug: Cyclophosphamide — together wit MTX and ASP in consolidation and together with cytarabine and 6-TG in reinduction
Drug: Cytarabine — part of different chemotherapy blocks in consolidation and reinduction
  Arms: Arm I intensification (cytarabine); Arm III reinduct.(doxorubicin hydrochl.); Arm IV reinduct.(daunorubicin hydrochl.)
Drug: Daunorubicin hydrochloride — part of induction and reinduction therapy
  Arms: Arm II intensification (clofarabine); Arm IV reinduct.(daunorubicin hydrochl.)
Drug: Dexamethasone — part of reinduction therapy
Drug: Doxorubicin hydrochloride — part of reinduction therapy
  Arms: Arm III reinduct.(doxorubicin hydrochl.)
Drug: Etoposide phosphate — part of different chemotherapy blocks
  Arms: Arm I intensification (cytarabine); Arm II intensification (clofarabine)
Drug: Mercaptopurine — part of different chemotherapy blocks
  Arms: Arm III reinduct.(doxorubicin hydrochl.); Arm IV reinduct.(daunorubicin hydrochl.)
Drug: Methotrexate — part of different chemotherapy blocks
Drug: Methylprednisolone — part of different chemotherapy blocks
  Arms: Arm I intensification (cytarabine); Arm II intensification (clofarabine)
Drug: Pegaspargase — part of different chemotherapy blocks
Drug: Thioguanine — part of different chemotherapy blocks
  Arms: Arm I intensification (cytarabine); Arm II intensification (clofarabine)
Drug: Vincristine sulfate — part of intravenous chemotherapy
Radiation: Whole-brain radiation therapy — patients with initial cns involvement receive cranial irradiation
  Arms: Arm I intensification (cytarabine); Arm II intensification (clofarabine)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than once drug (combination chemotherapy) may kill more cancer cells. Radiation therapy uses high-energy x-rays to kill cancer cells. It is not yet known whether giving clofarabine or high-dose cytarabine, pegaspargase, and combination chemotherapy followed by daunorubicin hydrochloride or doxorubicin hydrochloride is more effective in treating young patients with acute lymphoblastic leukemia.

PURPOSE: This randomized phase II/III trial is studying the side effects of giving clofarabine compared with giving high-dose cytarabine, pegaspargase, and combination chemotherapy followed by daunorubicin hydrochloride or doxorubicin hydrochloride and to see how well it works in treating young patients with T-cell acute lymphoblastic leukemia or precursor B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the safety and efficacy of clofarabine combined with pegaspargase in patients with high-risk acute lymphoblastic leukemia during the first phase of the study. (Phase II)
* To investigate, in terms of minimal-residual disease (MRD), the cytotoxic efficacy of clofarabine compared with high-dose cytarabine in combination with pegaspargase in these patients. (Phase III)
* To compare the incidence of infectious complications after the administration of daunorubicin hydrochloride versus doxorubicin hydrochloride during reinduction.

Secondary

* To compare the safety profiles of clofarabine and pegaspargase versus high-dose cytarabine and pegaspargase in these patients.
* To compare, in terms of MRD, the efficacy of clofarabine and pegaspargase and high-dose cytarabine and pegaspargase, respectively, versus methotrexate, cyclophosphamide, and asparaginase in study GER-COALL-07-03, the historical control group (retrospective comparison).
* To determine the influence of MRD-based stratification in COALL-09 on overall survival and event-free survival in a historical comparison of previous COALL studies.

OUTLINE: This is a multicenter, sequential phase II/III study. Patients are stratified to low risk (LR) or high risk (HR) depending on peripheral white blood cell count on diagnosis, age on diagnosis, and immunological subtype. Patients undergo 2 randomizations (1 during intensification and 1 during reinduction) in the study.

* Preliminary treatment: All patients receive daunorubicin hydrochloride IV over 24 hours on day -7 and methotrexate intrathecally (IT) once on day -9, -8, or -7.
* Induction: All patients receive vincristine IV on days 1, 8, 15, and 22; daunorubicin hydrochloride IV over 24 hours on days 1, 8, and 15; and oral prednisone 3-4 times daily on days 1-28.

Patients are assessed for minimal-residual disease (MRD) status after induction phase. Patients not in remission on day 29 are treated off study. Patients with LR disease are further stratified to LR-reduced (LR-R), LR-standard (LR-S), and LR-intensified (LR-I) groups; patients with HR disease are further stratified to HR-reduced (HR-R), HR-standard (HR-S), and HR-intensified (HR-I) groups. Patients in the LR-R and HR-R groups do not undergo randomization during study.

* Intensification (randomization 1): Patients receive therapy according to risk and disease subtypes. Some patients in different risk group are randomized* to receive high-dose (HD) cytarabine and pegaspargase or clofarabine and pegaspargase.

  * LR-R and LR-S: Patients receive medium-high-dose (mHD) methotrexate IV over 24 hours on days 50, 64, and 78; etoposide phosphate IV over 1-2 hours and cytarabine IV over 1 hour on day 66; oral mercaptopurine on days 50-56 and 78-120; oral thioguanine on days 64-70; and methotrexate IT on days 29, 50, 64, and 78. Patients in LR-S group who still have a detectable MRD load on day 29 are randomized (randomization 1) to 1 of 2 arms to receive cytarabine and pegaspargase vs. clofarabine and pegaspargase.

    * Arm I (cytarabine and pegaspargase) Patients receive HD cytarabine IV over 3 hours twice daily on days 29-31 and pegaspargase IV over 2 hours on days 31, 52, and 80.
    * Arm II (clofarabine and pegaspargase) Patients receive clofarabine IV over 2 hours on days 29-33 and pegaspargase IV over 2 hours on days 33, 52, and 80.
  * LR-I and precursor B-cell acute lymphoblastic leukemia (ALL) HR-S and HR-I: Patients receive cyclophosphamide IV over 30 minutes on days 50 and 64; mHD IV over 24 hours on days 51, 65, 78, and 92; etoposide phosphate IV over 1-2 hours and cytarabine IV over 1 hour on days 80 and 94; oral mercaptopurine on days 64-70 and 92-98; oral thioguanine on days 78-84; and methotrexate IT on days 29, 51, 65, 78, and 92. All precursor B-cell ALL patients with a detectable MRD load on day 29 and T-cell ALL patients with an MRD load ≥ 10³ on day 29 are randomized* (randomization 1) to 1 of 2 arms to receive cytarabine and pegaspargase vs. clofarabine and pegaspargase.

    * Arm I (cytarabine and pegaspargase) Patients receive HD cytarabine IV over 3 hours twice daily on days 29-31 and 106-108 and pegaspargase IV over 2 hours on days 31, 53, 67, and 108.
    * Arm II (clofarabine and pegaspargase) Patients receive clofarabine* IV over 2 hours on days 29-33 and pegaspargase IV over 2 hours on days 33, 53, 67, and 108.
  * NOTE: *In phase II, all patients with an MRD load of ≥ 104 (on day 29) receive clofarabine and pegaspargase without randomization.
  * T-cell ALL HR (HR-R, HR-S, and HR-I): Patients receive cyclophosphamide IV over 30 minutes on days 29 and 64; mHD methotrexate IV over 24 hours on days 30, 65, 78, and 92; etoposide phosphate IV over 1-2 hours and cytarabine IV over 1 hour on days 80 and 94; oral mercaptopurine on days 64-70 and 92-98; oral thioguanine on days 78-84; and methotrexate IT on days 30, 43, 65, 78, and 92. Patients in HR-S and HR-I group are randomized* (randomization 1) to 1 of 2 arms to receive cytarabine and pegaspargase vs. clofarabine and pegaspargase.

    * Arm I (cytarabine and pegaspargase): Patients receive HD cytarabine IV over 3 hours twice daily on days 43-45 and 106-108 and pegaspargase IV over 2 hours on days 32, 45, 67, and 108.
    * Arm II (clofarabine and pegaspargase): Patients receive clofarabine IV over 2 hours on days 43-47 and pegaspargase IV over 2 hours on days 32, 47, 67, and 108.

Patients in HR-I group also receive amsacrine IV over 4 hours and etoposide phosphate IV over 2 hours on days 127 and 128, methylprednisolone IV over 30 minutes on days 127-130, and methotrexate IT on day 127, at the end of intensification.

NOTE: *In phase II, all patients with an MRD load of ≥ 103 (on day 43) receive clofarabine and pegaspargase without randomization.

* CNS therapy: All patients with initial CNS involvement undergo cranial radiotherapy for a total of 12 or 18 Gy. HR patients (precursor B-cell ALL with initial WBC count ≥ 200/nL and T-cell ALL with initial WBC count ≥ 100/nL) with no initial CNS involvement also undergo cranial radiotherapy for a total of 12 Gy, beginning 2-3 weeks after the last dose of HD cytarabine or clofarabine. LR patients and HR patients (precursor B-cell ALL with initial WBC count < 200/nL and T-cell ALL with initial WBC count < 100/nL) with no initial CNS involvement do not receive initial cranial radiotherapy. At the beginning of CNS therapy, before cranial radiotherapy, HR-I patients receive vincristine IV on day 1; doxorubicin hydrochloride IV over 24 hours on day 1; oral dexamethasone 3 times daily on days 1-7; and pegaspargase IV over 2 hours on day 7.

All patients receive interim therapy comprising 3 doses (2 in week 1 and 1 in week 3) of methotrexate IT and oral mercaptopurine daily during the 4 weeks between intensification and reinduction.

* Reinduction (randomization 2): Patients undergo reinduction immediately after completion of interim therapy. Patients in LR-S, LR-I, HR-S, and HR-I groups are randomized to 1 of 2 arms (doxorubicin hydrochloride vs. daunorubicin hydrochloride)

  * LR-S: Patients receive vincristine IV on days 1 and 8, oral dexamethasone on days 1-14, pegaspargase IV over 2 hours on day 9, cyclophosphamide IV over 30 minutes on day 22, cytarabine IV or intramuscularly (IM) on days 23-26, oral thioguanine on days 22-28, and methotrexate IT on days 1, 22, and 36.

    * Arm III (doxorubicin hydrochloride) Patients receive doxorubicin hydrochloride IV over 24 hours on days 1 and 8.
    * Arm IV (daunorubicin hydrochloride): Patients receive daunorubicin hydrochloride IV over 24 hours on days 1 and 8.
  * LR-R and HR-R: Patients are not randomized. They receive vincristine IV on days 1 and 8, oral dexamethasone on days 1-14, pegaspargase IV over 2 hours on day 8, and methotrexate IT on days 1 and 15.
  * LR-I, HR-S, and HR-I: Patients receive vincristine IV on days 1, 8, 22, and 29; oral dexamethasone twice daily on days 1-14 and 22-35; cyclophosphamide IV over 30 minutes on days 43 and 57; cytarabine IV or IM on days 43-46 and 57-60; oral thioguanine on days 43-49 and 57-63; and methotrexate IT* on days 1, 22, and 43.

    * Arm III (doxorubicin hydrochloride) Patients receive doxorubicin hydrochloride IV over 24 hours on days 1, 8, 22, and 29.
    * Arm IV (daunorubicin hydrochloride) Patients receive daunorubicin hydrochloride IV over 24 hours on days 1, 8, 22, and 29.

NOTE: *Patients who underwent cranial radiotherapy do not receive methotrexate IT.

* Maintenance: Beginning 2-3 weeks after reinduction, all patients receive oral mercaptopurine daily and oral methotrexate weekly for 2 years. Except for LR-R and HR-R, patients also receive pegaspargase IV over 2 hours every 3 weeks for 3 doses. Patients who have not undergone CNS radiotherapy receive methotrexate IT at 3, 6, and 9 months.

Blood and bone marrow samples may be collected periodically for research studies.

After completion of study treatment, patients are followed monthly for 1 year, every 3 months for 2 years, every 6 months for 2 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 41 high-risk patients will be accrued for phase II, 296 patients for the first randomization (phase III), and 396 patients for the second randomization will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

diagnosis after the first and before the 18th birthday AND confirmed diagnosis of acute B-precursor or or T-cell leukemia AND parents or guardians/patients give consent for inclusion in the study and transmission of data AND if none of exclusion criteria is accomplished

Exclusion criteria:

BCR/ABL rearrangement positive OR prior cytostatic treatment lasting > 7 days or prior treatment with cytostatic drugs other than vincristine, daunorubicin and prednisone OR prior severe illnesses which make treatment per the protocol impossible from the outset (BUT trisomy 21 is not an exclusion criterion) OR absence of the baseline data required for assignment to a risk group in accordance with the protocol (BUT patients for whom the MRD value could not be determined for technical reasons will be treated as protocol patients) OR the disease is a secondary malignancy or relapse OR death before the start of treatment

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 745 (Actual)
Dates: Start 2010-10; Primary Completion 2019-12 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of clofarabine combined with pegaspargase (phase II) | at day 21 after chemotherapy
  minimal residual disease diagnostic, toxicity form

SECONDARY OUTCOMES:
Incidence of infectious complications after administration of daunorubicin hydrochloride vs doxorubicin hydrochloride | at the end of reinduction therapy
  toxicity form

CONTACTS AND LOCATIONS:
Overall Officials: Martin Horstmann, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (14):
- Germany (14):
  - Krankenanstalten Gilead gCmbH Neurochirurgische Klinik, Bielefeld
  - Klinikum Bremen-Mitte, Bremen
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Klinik und Poliklinik Fuer Kinder-und Jugendmedizin - Universitaetsklinikum Greifswald, Greifswald
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Klinikum Krefeld GmbH, Krefeld
  - Universitaets - Kinderklinik, Leipzig
  - Johannes Gutenberg University, Mainz
  - Dr. von Haunersches Kinderspital der Universitaet Muenchen, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinik St. Hedwig-Kinderklinik, Regensburg
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Helios Kliniken Wuppertal University Hospital, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trial summary from the information portal of the German Society of Paediatric Oncology and Haematology (GPOH) — https://www.kinderkrebsinfo.de/health_professionals/clinical_trials/pohkinderkrebsinfotherapiestudien/coall_08_09/index_eng.html